CLINICAL TRIAL: NCT02828540
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase II Clinical Trial to Assess the Efficacy and to Evaluate Safety of HT047 in Patients With Acute Ischemic Stroke
Brief Title: Clinical Trial to Assess the Efficacy and to Evaluate Safety of HT047 in Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hocheol Kim (Other)
Responsible Party: Sponsor-Investigator, Hocheol Kim, Professor, Kyunghee University
Organization: Kyunghee University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HT047-201
Record Dates: First submitted 2016-06-24; First posted 2016-07-11 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Ischemic Stroke
Keywords: HT047; Pueraria lobata; Scutellaria baicalensis
MeSH Terms: conditions — Ischemic Stroke | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HT047 High-dose group (Experimental): three times a day dosing schedule 3 tablets per dose
  Interventions: Drug: HT047 High-dose group
- HT047 Low-dose group (Experimental): three times a day dosing schedule 3 tablets per dose
  Interventions: Drug: HT047 Low-dose group
- Placebo (Placebo Comparator): three times a day dosing schedule 3 tablets per dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HT047 High-dose group — HT047 2250mg, three times a day dosing schedule, 3 tablets per dose
  Arms: HT047 High-dose group
Drug: HT047 Low-dose group — HT047 1500mg, three times a day dosing schedule, 3 tablets per dose
  Arms: HT047 Low-dose group
Drug: Placebo — placebo having the same appearance as HT047 Tab. 250mg
  Arms: Placebo

SUMMARY:
To assess the efficacy and to evaluate safety of HT047 in patients with acute ischemic stroke

DETAILED DESCRIPTION:
This clinical study is designed to initiate treatment with high or low dose HT047 or placebo in subjects with acute ischemic stroke within 2 weeks of onset of the disease and evaluate neurological function recovery in these subjects as measured by the extent of motor function recovery at Week 12 of treatment.

Subjects must have had a recent onset of acute ischemic stroke as confirmed by brain imaging. In terms of symptoms of ischemic stroke, patients who have motor function impairment with FMA motor score ≤ 55 as well as neurological function impairment with K-NIHSS score ≥ 4 and ≤ 15 are eligible for study participation. A subject who is considered by the investigator to be appropriate for study participation and provides informed consent will participate in this study.

At baseline, subjects will be randomized to HT047 high dose group (2250 mg/day), HT047 low dose group (1500 mg/day), or placebo group in a 1:1:1 ratio in a double blind fashion and be treated with the investigational product for 12 weeks starting from the next morning of baseline with a three times a day dosing schedule, 3 tablets per dose.

Since this is a first-in-human trial for HT047, subjects will have a study visit at Week 1 (Day 7) of participation for laboratory tests, ECG, and chest x-ray. A one-month portion of the investigational product will be supplied. During study treatment, subjects will visit the hospital at Weeks 1, 4, 8, and 12.

During the Week 1 visit, the above tests will be performed and the subject's physical status will be checked before he/she is sent home. In the subsequent visits, neurological function assessment and drug exchange will be carried out. At each visit, the study staff should carefully check the subject's medication compliance and verify the accurate number of remaining doses to be countered.

After 12 weeks of study conduct as shown in the above figure, at Week 12, laboratory tests performed at Week 1 will be repeated and overall change in the subject's status will be confirmed before all study procedures are ended.

ELIGIBILITY:
Inclusion Criteria:

1. Adult at the age of ≥ 19
2. Diagnosis of acute ischemic stroke by brain imaging within 14 days of screening
3. FMA motor score ≤ 55 with arm or leg weakness at screening
4. K-NIHSS score ≥ 4 and ≤ 15 at screening
5. Individuals who have visual and hearing abilities to perform the trial; who are able to understand the words and sentences necessary to evaluate the efficacy and safety, as well as the investigator's instructions; and who are able to communicate (such as gestures, writing, speaking, etc.)
6. Voluntary written informed consent to study participation

Exclusion Criteria:

1. Presence of motor function impairment, which is caused by previous stroke except acute ischemic stroke occurring within 14 days of screening (A subject with previous history of stroke may participate if he/she showed no motor function impairment and the K-mRS score was ≤1 (0-1))
2. Diagnosis of and current treatment for degenerative neurological diseases, e.g., Parkinson's disease and Alzheimer's disease
3. Current treatment with amphetamines, selective serotonin reuptake inhibitors, or antipsychotics
4. Presence of brain diseases, such as brain tumor, traumatic brain damage, arteriovenous malformation, or moyamoya disease, or ischemic stroke caused by these diseases
5. Impaired ability to walk upright due to other illness prior to screening
6. Unstable vital signs at screening based on the judgment of the investigator e.g., systolic blood pressure ≥ 170mmHg despite antihypertensive treatment or other symptoms such as hyperthermia, tachycardia, or hyperventilation
7. Diagnosis of liver diseases prior to screening, such as hepatitis and liver cirrhosis, or current treatment for these diseases
8. Continuous treatment with potentially hepatotoxic drugs e.g., current treatment with propylthiouracil, ketoconazole, isoniazid, valproic acid, phenytoin, etc. that may induce acute hepatotoxicity
9. Severe, New York Heart Association (NYHA) Class III or higher heart failure at screening [NYHA Classes of heart failure] Class I: patients with no limitation of activities; they suffer no symptoms from ordinary activities.

   Class II: patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion.

   Class III: patients with marked limitation of activity; they are comfortable only at rest.

   Class IV: patients who should be at complete rest, confined to bed or chair; any physical activity brings on.
10. Diagnosis of or treatment for cancer within 6 months of screening or presence of recurrent or metastatic cancer
11. Treatment with or intake of traditional oriental medicine (herbal medicine) or health functional foods containing potentially hepatotoxic plants, such as Germander (Teucrium chamaedrys, Teucrium polium), toothed clubmoss (Lycopodium serratum), or celandine (Chelidonium majus), within 4 weeks prior to study participation
12. Treatment with or intake of traditional Korean medicine containing pueraria root and/or scutellaria root or other drugs or health functional foods containing their respective index components, i.e. puerarin and baicalin, within 4 weeks prior to study participation
13. Hematologic findings as follows

    ① Increased serum aspartate or alanine aminotransferase (AST/ALT) levels ≥ 1.5 x site specific upper limit of normal in laboratory test

    ② Decreased hemoglobin (Hb) level (Hb< 10 g/dl), decreased platelet (PLT) level (PLT< 100,000/mm3), or hematocrit (Hct) level < 25% in whole blood count test.

    ③ Increased serum creatinine (Cr) level (Cr > 2.0 mg/dl) in laboratory test or patient on dialysis
14. Pregnant or lactating women A woman of childbearing potential can participate in the study only if non-pregnancy is confirmed.

    Subjects must use a double barrier method or must have been surgically sterilized.
15. Previous participation in a clinical study for another drug within 3 months of screening. A subject who participated in an observational study that did not involve drug treatment may participate in this study.
16. Individuals who are considered by the investigator to be inadequate for study participation due to other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-08-04; Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Change at Week 12 of treatment with HT047 Tab. from baseline in Korean version of Fugl-Meyer Assessment (FMA) motor function score | 12 weeks
  Total score of motor function test for upper extremity in 66 marks plus total score of motor function test for lower extremity in 34 marks is 100 marks.

SECONDARY OUTCOMES:
Change at Weeks 4, 8 and 12 from baseline in FMA motor function score | 4weeks, 8weeks, 12 weeks
  Total score of motor function test for upper extremity in 66 marks plus total score of motor function test for lower extremity in 34 marks is 100 marks.
Change at Weeks 4, 8, and 12 from baseline in FMA motor function score according to the timing of treatment initiation after the onset of stroke. | 4weeks, 8weeks, 12 weeks
  Total score of motor function test for upper extremity in 66 marks plus total score of motor function test for lower extremity in 34 marks is 100 marks.
Change at Weeks 4, 8, and 12 from baseline in FMA motor function score according to the presence of prognostic risk factors (hypertension, diabetes, dyslipidemia, etc.) | 4weeks, 8weeks, 12 weeks
  Total score of motor function test for upper extremity in 66 marks plus total score of motor function test for lower extremity in 34 marks is 100 marks.
Change at Weeks 4 and 12 from baseline in Korean-National Institutes of Health Stroke Scale (K-NIHSS) scores | 4weeks, 12 weeks
  Total score of K-NIHSS would be scored by 11 categories.
Change at Weeks 4 and 12 from baseline in Korean modified Rankin Scale (K-mRS) scores | 4weeks, 12weeks
  Different 6 questions can be scored by 0-5 marks.
Proportion of subjects with K-NIHSS score 0 - 2 at Week 12 | 12weeks
  Total score of K-NIHSS would be scored by 11 categories.
Proportion of subjects with K-mRS score 0, ≤ 1, and ≤ 2 at Week 12 | 12weeks
  Different 6 questions can be scored by 0-5 marks.
Change at Weeks 4 and 12 from baseline in Korean Modified Barthel Index (K-MBI) score | 4weeks, 12weeks
  Total scores (0-100) should be rated by 5 stages in 10 categories.

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Il Chang, Principal Investigator — Kyung Hee University Hospital
Locations (8):
- South Korea (8):
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - Chosun University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Hanyang University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heo SH, Song J, Kim BJ, Kim H, Chang DI; HT047 investigators. Rationale and design to assess the efficacy and safety of HT047 in patients with acute ischemic stroke: A multicenter, randomized, double-blind, placebo-controlled, parallel-group, phase II trial. Medicine (Baltimore). 2019 Oct;98(43):e17655. doi: 10.1097/MD.0000000000017655. PMID 31651889